CLINICAL TRIAL: NCT02835547
Title: Evaluation and Management of Cardiovascular Risk Factors in Inflammatory and Acquired Dysimmune Diseases (CARMIN)
Acronym: CARMIN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50841
Record Dates: First submitted 2016-06-21; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Inflammatory and Acquired Dysimmune Diseases
Keywords: cardiovascular event; risk factors; inflammatory diseases and acquired dysimmune
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Systemic lupus erythematosus: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection
- Rheumatoid arthritis: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection
- Psoriasis: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection
- Scleroderma: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection
- Hematopoietic stem cells transplants: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection
- Kidney transplants: Data collection of risk factors (collected retrospectively - 5 years) and cardiovascular events (collected prospectively - 2 years).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Risk factors will be collected retrospectively (5 years) and cardiovascular events prospectively (2 years)

SUMMARY:
The hypothesis is that chronic inflammatory dysimmune state promotes the development of cardiovascular complications. The biological assumption is based on the fact that chronic inflammation promotes lesions of the vessel wall (endothelial alterations, calcification, atherosclerosis). The clinical aim is to allow to identify high-risk patients and to act in prevention.

The project CARMIN involves the assessment of cardiovascular risk factors, their management, and their influence on cardiovascular prognosis in patients with autoimmune diseases and immunodeficiencies acquired. It is based on the creation and monitoring of a cohort of patients with different types of dysimmune disorders: systemic lupus erythematosus, rheumatoid arthritis, psoriasis, scleroderma, systemic vasculitis ANCA, kidney transplants, and hematopoietic stem cells transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the various services of medical specialties pole of the Edouard Herriot hospital
* The diagnosis of the pathology selected for this study based on a clear clinical and biological evaluation supported by criteria specific to each pathology and compatible with international standards.
* Date of diagnosis should not be less than 5 years (+/- 1 year), except for scleroderma patients where it has been extended to 10 years.
* For kidney transplant patients the investigators take into account only patients with a maximum of 2 years of dialysis before graft.

Exclusion Criteria:

* Diabetic patients
* HIV seropositive
* Patients with multiple pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus, rheumatoid arthritis, psoriasis, scleroderma, kidney transplants, or hematopoietic stem cells transplants
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The occurrence of any cardiovascular event (will be recorded from the patient files and/or phone calls to patient") | 2 years
  The cardiovascular events : cardiovascular death, myocardial infarction, stroke, peripheral arterial disease, ischemic manifestations in other territories, heart failure, arrhythmia, deep vein thrombosis or pulmonary embolism.